CLINICAL TRIAL: NCT07027774
Title: A Multicenter, Prospective, Randomized, Controlled Study Evaluating the Progression of Renal Function in Patients With Late-Stage Chronic Kidney Disease Treated With Henagliflozin
Brief Title: Effect of Henagliflozin on Renal Outcomes in Non-dialysis Patients With Advanced Chronic Kidney Disease : A Multicenter Prospective, Randomized Controlled Trial（HERO -aCKD）
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAW2024104
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease Stage 4
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — henagliflozin; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Henagliflozin 5mg Group (Experimental): Henagliflozin 5 mg once daily + RAASi-based comprehensive strategy (optional)
  Interventions: Drug: Henagliflozin 5 mg Group
- Henagliflozin 10mg Group (Experimental): Henagliflozin 10 mg once daily + RAASi-based comprehensive strategy (optional)
  Interventions: Drug: Henagliflozin 10 mg Group
- Conventional therapy group (Active Comparator): RAASi-based comprehensive strategy (e.g., ramipril + lipid control + glycemic management)
  Interventions: Drug: Conventional therapy group

INTERVENTIONS:
Drug: Henagliflozin 5 mg Group — Henagliflozin 5 mg once daily plus KDIGO-based comprehensive management strategy (e.g., RAAS inhibitors）
  Arms: Henagliflozin 5mg Group
Drug: Henagliflozin 10 mg Group — Henagliflozin 10 mg once daily plus KDIGO-based comprehensive management strategy (e.g., RAAS inhibitors）
  Arms: Henagliflozin 10mg Group
Drug: Conventional therapy group — KDIGO-based comprehensive management strategy (e.g., RAAS inhibitors）
  Arms: Conventional therapy group

SUMMARY:
This is a multicenter, prospective, randomized, controlled study that will enroll approximately 429 subjects. The screening period will last 4-8 weeks. Subjects will undergo pre-screening based on eGFR and urinary albumin-to-creatinine ratio (UACR). Only non-dialysis subjects meeting the following criteria confirmed by local laboratories within 6 months prior to screening will be eligible for central laboratory screening:

10 mL/min/1.73m² ≤ eGFR < 30 mL/min/1.73m² and 150 mg/g (16.95 mg/mmol) ≤ UACR < 5000 mg/g (565 mg/mmol).

Unless contraindicated due to intolerance, subjects with 20 mL/min/1.73m² ≤ eGFR < 30 mL/min/1.73m² must receive stable, maximally tolerated labeled daily doses of ACEi or ARB for at least 4 weeks prior to randomization. For subjects with 10 mL/min/1.73m² ≤ eGFR < 20 mL/min/1.73m², investigators will determine ACEi/ARB treatment based on patient condition per KDIGO guidelines. Other antihypertensive, lipid-lowering, and glucose-lowering therapies should be stabilized for approximately 4 weeks before randomization. Investigators are encouraged to maintain stability of medications known to affect serum creatinine levels during screening and approximately 2 weeks prior to any serum chemistry measurements throughout the study. Eligible subjects will be randomized in a 1:1:1 ratio to receive Henagliflozin (10 mg q.d., 5 mg q.d.) or conventional therapy.

Thereafter, subjects will undergo laboratory assessments, concomitant medication review, adverse event collection, and clinical endpoint ascertainment at Week 4 (Day 30), Week 12 (Day 90), and Week 24 (Day 180), followed by every 12-week intervals. Throughout the study, all subjects will receive glycemic, blood pressure (target SBP <140 mmHg and DBP <90 mmHg), and lipid management according to current guidelines. All subjects will complete an end-of-study visit. Subjects discontinuing study drug prematurely should continue all subsequent study visits.

ELIGIBILITY:
Inclusion Criteria:

* The investigator considers that the participant does not require Henagliflozin or any other SGLT-2 inhibitor therapy, nor deems such therapy absolutely inappropriate; and based on local laboratory results within 6 months before the screening visit and at the screening visit, the following criteria must be met:

  1. 10 mL/min/1.73m² ≤ eGFR < 30 mL/min/1.73m² (CKD-EPI equation), and
  2. 150 mg/g (16.95 mg/mmol) ≤ Urine Albumin-to-Creatinine Ratio (UACR) < 5000 mg/g (565 mg/mmol)
* Age ≥ 18 years, male or femal
* Participants with 20 mL/min/1.73m² ≤ eGFR < 30 mL/min/1.73m² must be on a stable and tolerated dose of an ACE inhibitor (ACEI) or ARB for at least 4 weeks, unless intolerant (reasons for intolerance must be documented). Participants with 10 mL/min/1.73m² ≤ eGFR < 20 mL/min/1.73m² should have ACEI/ARB use determined by the investigator based on the patient's clinical status and KDIGO guideline recommendations;
* Anticipated time to requiring dialysis is greater than 1 month;
* Provision of written informed consent (illiterate participants may use a thumbprint in lieu of a signature).

Exclusion Criteria:

* Received SGLT2 inhibitor treatment within 8 weeks prior to enrollment or with a history of SGLT2 inhibitor intolerance;
* Receiving combined therapy with an ACE inhibitor (ACEi) and an ARB, or a renin inhibitor combined with ACEi or ARB (based on self-report at screening and randomization visits);
* On maintenance dialysis, has a functioning kidney transplant, or is a planned living donor transplant recipient (based on self-report at screening and randomization visits);
* Polycystic kidney disease, active lupus nephritis, or systemic vasculitis;(5) Symptomatic hypotension, or systolic blood pressure <90 mmHg or >180 mmHg at screening;
* ALT or AST levels >3 times the upper limit of normal (ULN) at screening;
* Received any intravenous immunosuppressive therapy within the previous 3 months; or any subject who received prednisone >45 mg/day (or equivalent dose) within the previous 3 months;
* Current use or use within 12 weeks prior to enrollment of glucagon-like peptide-1 (GLP-1) receptor agonist medications (e.g., liraglutide, semaglutide, dulaglutide, etc.) or current participation in another clinical trial of glucose-lowering drugs that may affect kidney or cardiovascular outcomes;(9) Severe malnutrition (serum albumin <25 g/L) and/or severe anemia (hemoglobin <70 g/L);
* Known poor adherence to clinical follow-up or medication;
* Myocardial infarction, unstable angina, or stroke within 12 weeks prior to enrollment;
* Underwent coronary revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass grafting [CABG]) or valve repair/replacement within 12 weeks prior to enrollment, or plans to undergo any of these procedures after randomization;(13) Any disease other than kidney or cardiovascular disease (e.g., but not limited to, malignancy) that, in the investigator's clinical judgment, is associated with a life expectancy of less than 2 years;
* Active malignancy requiring treatment at the time of the first visit (except for successfully treated basal cell carcinoma, treated squamous cell carcinoma, or thyroid cancer);
* Currently pregnant, breastfeeding, or a woman of childbearing potential (WOCBP) unless using a highly effective method of contraception;
* Type 1 diabetes;(17) Investigator considers the patient unable to understand and/or comply with the study procedures and/or follow-up, or any condition that, in the investigator's opinion, may lead to the patient's inability to complete the study.
* Additionally, subjects will be excluded at the randomization visit if any of the following occur:

  1. Did not adhere to the run-in treatment;
  2. No longer willing to be randomized and followed for at least 2 years;
  3. Considered unsuitable for randomization by the local investigator; OR experienced ketoacidosis, heart attack (myocardial infarction), stroke, hospitalization for heart failure, hospitalization for urinary tract infection, or acute kidney injury during the run-in period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
eGFR total slope change from 4 to 52 weeks | 52 weeks

SECONDARY OUTCOMES:
Total eGFR slope at 1 year post-randomization | 56 weeks
Composite endpoint of kidney disease progression ，hospitalization for heart failure, or cardiovascular death. | 56 weeks
  Composite endpoint of kidney disease progression (defined as a sustained decline in eGFR of ≥40% from baseline, sustained eGFR <7.5 mL/min/1.73m², initiation of maintenance dialysis or kidney transplantation, or kidney death), hospitalization for heart failure, or cardiovascular death.
Kidney disease progression (sustained eGFR decline ≥40%, sustained eGFR <7.5 mL/min/1.73m², initiation of maintenance dialysis or kidney transplantation, or kidney death). | 56 weeks
  Kidney disease progression is defined as a sustained decline in eGFR of ≥40% from baseline since randomization, sustained decline in eGFR to <7.5 mL/min/1.73m², initiation of maintenance dialysis or kidney transplantation, or death due to kidney disease.
Composite endpoint of major adverse cardiovascular events (MACE) (defined as cardiovascular death, myocardial infarction, stroke, or hospitalization for heart failure) | 56 weeks
Composite endpoint of initiation of maintenance dialysis or kidney transplantation, kidney death, or cardiovascular death. | 56 weeks
Composite endpoint of initiation of maintenance dialysis, kidney transplantation, or kidney death. | 56 weeks
Composite endpoint of cardiovascular death, myocardial infarction, stroke, hospitalization for heart failure, or unstable angina. | 56 weeks
Cardiovascular death or hospitalization for heart failure. | 56 weeks
All-cause hospitalization | 56 weeks

IPD SHARING:
Plan to Share IPD: No